CLINICAL TRIAL: NCT06253494
Title: Pembrolizumab, Lenvatinib and IL-15 Superagonist N-803 in Combination With HER2 Targeting Autologous Dendritic Cell (AdHER2DC) Vaccine in Participants With Advanced or Metastatic Endometrial Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10001557; 001557-C
Record Dates: First submitted 2024-02-09; First posted 2024-02-12 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11-25

CONDITIONS: Endometrial Cancer; Cancer of Endometrium; Carcinoma of Endometrium; Endometrial Carcinoma
Keywords: Cancer Vaccine; Combination of anti-cancer drugs; Immunotherapy; HER2 Positive Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — pembrolizumab; ALT-803; lenvatinib; Biological Assay

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): AdHER2DC vaccine + pembrolizumab + de-escalating doses of lenvatinib
  Interventions: Biological: AdHER2DC vaccine; Biological: Pembrolizumab; Drug: Lenvatinib; Device: PATHWAY HER2 (4B5) assay
- Arm 2 (Experimental): AdHER2DC vaccine + N-803 + pembrolizumab + RP2D of lenvatinib
  Interventions: Biological: AdHER2DC vaccine; Biological: Pembrolizumab; Biological: N-803; Drug: Lenvatinib; Device: PATHWAY HER2 (4B5) assay

INTERVENTIONS:
Biological: AdHER2DC vaccine — AdHER2DC vaccine is given by intradermal injections on Day 1 of cycles 1-3 (priming) followed by optional boost doses (up to 3), on Day 1 of cycles 6, 9, 12
Biological: Pembrolizumab — Pembrolizumab is given by IV infusion on Day 8 of cycle 1 and Day 1 of cycles 2-16
Biological: N-803 — N-803 is given by subcutaneous injections on Day 1 of cycles 1-16
  Arms: Arm 2
Drug: Lenvatinib — Lenvatinib is taken orally on Days 8-28 on cycle 1 and every day of cycles 2-16
Device: PATHWAY HER2 (4B5) assay — Used during screening to estimate eligibility

SUMMARY:
Background:

Endometrial cancer (EC) of the uterus is becoming more common in the US. Sometimes EC often has increased levels of a protein called HER2. Cancers with HER2 tend to be more aggressive and have poorer outcomes.

Objective:

To test 2 study drugs-a vaccine that targets HER2 (AdHER2DC) plus a drug that supercharges immune cells that kill tumor cells (N-803)-combined with 2 FDA-approved cancer treatment drugs in people with EC.

Eligibility:

Adults aged 18 and older with HER2-positive EC that returned or got worse after treatment.

Design:

AdHER2DC vaccine is made from each participant s own blood. Participants will undergo apheresis: Blood is removed from the body through a tube attached to a needle. The blood passes through a machine that separates out the target cells. The remaining blood is returned to the body through a second needle. A special catheter may be needed.

The first treatment cycle is 28 days; each cycle after that will be 21 days.

All participants will get the 2 approved drugs and the vaccine. One drug is a tablet taken by mouth once a day, every day. The other drug is given through a tube attached to a needle inserted into a vein.

The vaccine is injected under the skin. Participants will receive the vaccine on day 1 of cycles 1, 2, and 3. Additional doses up to 3 doses will be give if possible.

Some participants will receive N-803. This drug is injected under the skin of the abdomen on day 1 of each cycle.

Treatment may last up to 1 year. Follow-up visits will continue up to 2 more years.

DETAILED DESCRIPTION:
BACKGROUND:

* Endometrial cancer (EC) is the most common gynecologic cancer in the US and the incidence peaks around 50-60 years of age. 5-year overall survival in patients with metastasis is around 20 percent and treatment after the second-line treatment has not been effective for long-term control.
* Pembrolizumab is approved for microsatellite instability (MSI)-high endometrial cancer which is rare.
* Pembrolizumab and lenvatinib combination therapy as second-line therapy in patients with advanced or metastatic EC showed promising antitumor activity. Recently, the Food and Drug Administration (FDA) approved pembrolizumab and lenvatinib in patients with advanced endometrial cancer who received prior chemotherapy after decades of lapse in adding new treatment options with an improved progression free survival (PFS) 6.6 months (vs 3.8 months in standard care chemotherapy), overall response rate 30 percent and median duration of response of 9.2 months.
* HER2 is positive in 30 percent of endometrial cancer and anti-HER2 therapy has shown clinical benefit in metastatic EC. Trastuzumab is used off-label with chemotherapy and as maintenance.
* An autologous dendritic cell vaccine that is transduced with an adenoviral vector expressing extracellular domain and transmembrane domain of HER2 (AdHER2DC vaccine) was well tolerated and showed a preliminary clinical benefit of 33.3 percent among 21 evaluable patients (NCT01730118, total enrolled n=33). No cardiotoxicity was noted. Immunogenicity analysis in a limited number of patients suggested induction of both humoral and cellular immune responses.
* The combination of pembrolizumab and lenvatinib in EC showed antitumor activity with manageable toxicity but still showed the responses in a limited group of patients. To overcome the resistance to immune checkpoint inhibitors, the combination regimen to induce the antitumor immune response by the AdHER2 vaccine, control the negative immune regulators and hostile tumor microenvironment by vascular endothelial growth factor (VEGF) inhibitor lenvatinib, and an immune stimulatory cytokine IL-15 superagonist N-803 has the potential to make the tumor more responsive to the immunotherapy creating mutual synergy.

OBJECTIVES:

* Phase I: To estimate recommended Phase II dose (RP2D) of pembrolizumab, lenvatinib, N-803, and AdHER2DC vaccine in participants with HER2 positive endometrial cancer
* Phase II: To preliminarily assess the efficacy of a combination of pembrolizumab, lenvatinib, N-803, and AdHER2DC vaccine in participants with HER2 positive endometrial cancer as determined by the proportion of participants without progression at 6 months

ELIGIBILITY CRITERIA:

* Age >=18 years.
* Metastatic or locally advanced endometrial cancer with HER2 immunohistochemistry (IHC) 1+, 2+ or 3+.
* Progressed after at least 1 line of standard of care (SOC) systemic therapy Participants may have received any number of prior cytotoxic agents.
* ECOG performance status <=2 and adequate organ function.

DESIGN:

* An open-label, two-arm, phase I/II study of pembrolizumab, lenvatinib, N-803, and AdHER2.
* During Phase I, we will estimate recommended Phase II dose (RP2D) of the lenvatinib in combination with AdHER2DC vaccine, pembrolizumab, and N-803.
* During Phase II we will continue to evaluate the safety and examine the efficacy of the study regimen at the RP2D of the lenvatinib in combination with AdHER2 DC vaccine, pembrolizumab, and N-803.
* Participants will undergo apheresis, and AdHER2DC vaccine will be generated by transducing the participants monocyte-derived dendritic cells with AdHER2 vector.
* Treatment will be delivered for up to 1 year or until progression or unacceptable toxicity.
* Up to 27 participants will be treated on this trial.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Histologically confirmed endometrial cancer.
* Radiographically confirmed metastatic or locally advanced disease.
* Evaluable (measurable or non-measurable) disease, per RECIST 1.1.
* HER2 IHC 1+, 2+ or 3+ tumor confirmed by PATHWAY HER2 (4B5) test. NOTE: The HER2 status in participants who had prior anti-HER2 therapy should be confirmed in the tumor tissue obtained after completing the anti-HER2 therapy.
* Participants must have received and progressed after at least one (1) line of systemic therapy for endometrial cancer.
* Age >=18 years.
* ECOG performance status <=2.
* Participants must have available tumor tissue or be willing to undergo a mandatory research biopsy. NOTE: Samples must be collected after HER2 directed therapy if the participant had anti-HER2 therapy.
* Participants must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count (ANC) > 1,000/microliter
  * Platelets > 100,000/microliter
  * Hemoglobin (Hgb) > 9 g/dL (any number of transfusions within 60 days before apheresis is allowed)
  * Total bilirubin <=1.5 X upper limit of normal (ULN). NOTE: In participants with Gilbert s Syndrome or known liver metastasis, total bilirubin <=3.0 X ULN is allowed
  * Aspartate aminotransferase (AST) / Alanine aminotransferase (ALT) <=3.0 X ULN. NOTE: AST/ALT <=5.0 X ULN is allowed in participants with known liver metastasis
  * An estimated creatinine clearance (CrCl) <=1.5 X ULN OR >30 mL/min/1.73 m2 for participants with creatinine levels >1.5 X ULN (calculated creatinine clearance (CrCl) (eGFR may also be used in place of CrCl)
  * Dip stick urine protein < 3 or urine protein < 1 gram (g)/24 hour if dip stick urine is >= 3+
* Hepatitis B virus (HBV)-infected participants can be enrolled if HBV DNA is undetectable. Hepatitis C virus (HCV)-infected participants can be enrolled if HCV RNA level is undetectable.
* Participants with previously treated non-active brain metastases or central nervous system metastases more than 28 days from definitive radiotherapy or surgery are eligible.
* Individuals of child-bearing potential (IOCBP) must agree to use highly effective contraception (hormonal, intrauterine device (IUD), tube ligation, a partner has had the previous vasectomy, abstinence) at the time of study entry, for the duration of study treatment, and up to 6 months after the last dose of the study drug(s).
* Nursing participants must be willing to discontinue nursing from study treatment initiation through 6 months after the last dose of the study drug(s).
* Participants must be able to understand and be willing to sign a written informed consent document.

EXCLUSION CRITERIA

* Administration of any standard of care or investigational checkpoint inhibitors (e.g., anti-CTLA, anti-PD-1, anti-PD-L1, anti-TIGIT, anti-TIM3, or anti-LAG3 antibodies or small molecules) within 6 months prior to apheresis.
* History of grade 3 or 4 immune related adverse events from the use of immune checkpoint inhibitors.
* History of Lenvatinib use
* History of severe immediate hypersensitivity reaction to compounds similar to study drugs or their components (e.g., monoclonal antibody preparations).
* Surgery to abdomen/pelvis/chest within 3 months prior to apheresis.
* Other malignancies diagnosed within 24 months prior to apheresis. NOTE: Participants who completed treatment for in-situ carcinomas (e.g., breast, cervix, bladder), or basal or squamous cell carcinoma of the skin are eligible if no ongoing treatment is needed per Standard of Care.
* Arterial or venous thromboembolism within 6 months prior to apheresis.
* History of cerebrovascular accident or stroke (transient ischemic attack, hemorrhagic or ischemic) within 6 months prior to apheresis.
* Functional or objective cardiac dysfunction: New York Heart Association (NYHA) Functional Capacity III or IV or Objective Assessment C or D.
* Fridericia's corrected QT interval (QTcF) >= 480 msec or evidence of third-degree AV block on screening electrocardiogram (ECG).
* Ejection fraction by screening echocardiogram < 50 percent.
* Participants requiring therapeutic anticoagulation regimen(s) (e.g., warfarin, rivaroxaban, apixaban, dabigatran, edoxaban, low molecular weight heparin [e.g., enoxaparin, dalteparin, tinzaparin], heparin, fondaparinux).
* History of gastrointestinal or non-gastrointestinal fistula >= Grade 3 (CTCAE v.5.0).
* Radiographic evidence of major blood vessel invasion/infiltration.
* History of hemoptysis or tumor bleeding within 1 month prior to apheresis.
* Current gastrointestinal malabsorption, gastrointestinal anastomosis, or any other condition that might affect the absorption of lenvatinib.
* Any form of primary immunodeficiency.
* Participants with active autoimmune disease or a history of autoimmune disease, which require immune suppressive treatment such as systemic corticosteroids or other systemic immune suppressants (e.g., methotrexate, cyclosporine, and biologics). NOTE: Participants with vitiligo, endocrine deficiencies on replacement dose are eligible.
* Systemic corticosteroid therapy of higher than a physiologic dose (the equivalent of prednisone 10 mg/day) within 14 days prior to apheresis. NOTE: Any topical steroid medications (e.g., corticosteroid creams, ointments, and eye drops) are allowed.
* Solid organ or allogeneic hematopoietic stem cell transplant recipients.
* Human immunodeficiency virus (HIV)-positive participants.
* Pregnancy (confirmed with beta-Human chorionic gonadotropin (HCG) serum or urine pregnancy test performed in IOCBP at screening).
* Uncontrolled intercurrent illness or situation that would limit compliance with study requirements.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase I: Estimate recommended RP2D of pembrolizumab, lenvatinib, N-803, and AdHER2DC vaccine in participants with HER2 positive endometrial cancer | Days 1-28 of Cycle 1
  Number of Dose Limiting Toxicities (DLT).
Phase II: Preliminarily assess the efficacy of a combination of pembrolizumab, lenvatinib, N-803, and AdHER2DC vaccine in participants with HER2 positive endometrial cancer | 6 months
  Defined as the time from the start of treatment to time of progression, death, or 6 months. The fraction who can be alive without progression at 6 months will be reported along with an 80% two-sided confidence interval (the lower bound is the one-sided 90% bound, which will be used to compare to an estimated 54-55% from the Makker 2022 result) and a 95% two-sided confidence interval.

SECONDARY OUTCOMES:
Determine the safety of the combination of pembrolizumab, lenvatinib, N-803, and AdHER2DC vaccine in participants with HER2 positive endometrial cancer | While on treatment (up to 1 year) and at the Safety Follow Up visit (30 days after treatment completion).
  For participants receiving 4 agents, their safety will be evaluated with respect to the grades and types of toxicities obtained. The results will be presented descriptively and tabled if appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Hoyoung M Maeng, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGap.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. Genomic data are made available via gbGaP through requests to the data custodians.

REFERENCES:
- [Background] Konecny GE, Santos L, Winterhoff B, Hatmal M, Keeney GL, Mariani A, Jones M, Neuper C, Thomas B, Muderspach L, Riehle D, Wang HJ, Dowdy S, Podratz KC, Press MF. HER2 gene amplification and EGFR expression in a large cohort of surgically staged patients with nonendometrioid (type II) endometrial cancer. Br J Cancer. 2009 Jan 13;100(1):89-95. doi: 10.1038/sj.bjc.6604814. Epub 2008 Dec 16. PMID 19088718
- [Background] Makker V, Colombo N, Casado Herraez A, Santin AD, Colomba E, Miller DS, Fujiwara K, Pignata S, Baron-Hay S, Ray-Coquard I, Shapira-Frommer R, Ushijima K, Sakata J, Yonemori K, Kim YM, Guerra EM, Sanli UA, McCormack MM, Smith AD, Keefe S, Bird S, Dutta L, Orlowski RJ, Lorusso D; Study 309-KEYNOTE-775 Investigators. Lenvatinib plus Pembrolizumab for Advanced Endometrial Cancer. N Engl J Med. 2022 Feb 3;386(5):437-448. doi: 10.1056/NEJMoa2108330. Epub 2022 Jan 19. PMID 35045221
- [Background] Constantine GD, Kessler G, Graham S, Goldstein SR. Increased Incidence of Endometrial Cancer Following the Women's Health Initiative: An Assessment of Risk Factors. J Womens Health (Larchmt). 2019 Feb;28(2):237-243. doi: 10.1089/jwh.2018.6956. Epub 2018 Nov 28. PMID 30484734
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001557-C.html